CLINICAL TRIAL: NCT01988571
Title: Preventing Anthracycline Cardiovascular Toxicity With Statins (PREVENT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00038639; U10CA081851 (NIH); 1R01HL118740-01 (NIH); REBACCCWFU 98213 (Other: NCI); NCI-2013-01760 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-11-01; First posted 2013-11-20 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Lymphoma
Keywords: Stage I breast cancer; Stage II breast cancer; Stage III breast cancer; Stage I Lymphoma; Stage II Lymphoma; Stage III Lymphoma; Stage IV Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Lymphoma | interventions — Atorvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Atorvastatin (Active Comparator): One 40 mg Atorvastatin tablet each morning by mouth for 24 months
  Interventions: Drug: Atorvastatin
- Arm 2 - Placebo (Placebo Comparator): One placebo tablet each morning by mouth for 24 months.
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 40 mg tablet taken by mouth each morning for 24 months.
  Other Names: Lipitor
Drug: Placebo — One placebo tablet taken each morning orally for 24 months.
  Other Names: sugar pill
  Arms: Arm 2 - Placebo

SUMMARY:
The purpose of this research study is to see if Atorvastatin (Lipitor) 40 mg by mouth daily decreases the chance of developing heart problems in individuals receiving adjuvant anthracycline-based chemotherapy for breast cancer of lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Specific Aim 1:

To determine if Atorvastatin(Lipitor) administration preserves left ventricular ejection fraction (LVEF) 24 months after initiation of Anthracycline-based adjuvant therapy for adjuvant treatment of breast cancer or lymphoma.

Specific Aim 2:

To determine if baseline to 6-month differences in LVEF predict baseline to 24-month differences in LVEF after Anthracycline-based adjuvant therapy and concomitant atorvastatin therapy.

To achieve these aims, we will perform a double-blind, placebo-controlled, randomized clinical trial of 0 or 40 mg of atorvastatin/day in 278 individuals scheduled to receive Anthracycline-based chemotherapy for treatment of Stage I-III breast cancer or lymphoma Stage I-IV with a projected > 2 year life expectancy. We will use innovative noninvasive magnetic resonance imaging (MRI) procedures to accurately measure LVEF. In addition, we will measure left ventricle (LV) volumes, myocardial strain, fibrosis, aortic pulse wave velocity (PWV) and wall thickness, all factors that can influence LVEF by altering LV pre-load, after-load, and contractility.19,20 Advanced serum biomarkers will be measured that assess for the presence of oxidative/nitrosative stress, systemic inflammation and circulating neurohormones that also may influence LVEF.

This study will test a new clinical paradigm to manage breast cancer: primary prevention of Anthracycline-based adjuvant therapy-related LV dysfunction using pre-treatment with low-cost statins. In addition, this trial will be the first systematic collection of data regarding the mechanism(s) and time course by which LV dysfunction and subsequent chronic heart failure (CHF) evolve in individuals given Anthracycline-based chemotherapy for breast cancer or lymphoma. These data will be useful to physicians trying to determine the optimal cardiac protection strategies when administering adjuvant chemotherapeutic regimens to their breast cancer or lymphoma patients. The objective of this research is to use inexpensive medications to preserve cardiovascular (CV) health and thereby improve overall survival in the growing number of breast cancer and lymphoma patients.

SECONDARY OBJECTIVES

Specific Aim 1:

To document the effect of Atorvastatin (Lipitor) on cognitive function using a battery of neurocognitive tests (HVLT, Rey-osterrieth Figure, controlled oral word association test (COWA), Trail-making Parts A and B, Digit Span and Grooved Pegboard) in breast cancer and lymphoma patients receiving an anthracycline.

Specific Aim 2:

To document the effect of Atorvastatin(Lipitor) on self-reported quality of life using validated questionnaires (PROMIS including: General form, Cog Concerns, Cog Abilities, Fatigue, Pain intensity and interference, Sleep Disturbance, Physical Functioning and Social Functioning) in breast cancer and lymphoma patients receiving an anthracycline.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer (including inflammatory and newly diagnosed recurrent breast cancer) or lymphoma Stage I-IV. (Patients should have a > 2 year life expectancy)
* Scheduled to receive adjuvant chemotherapy with an Anthracycline (doxorubicin and epirubicin)
* 21 years of age or older
* LVEF > 50% (Most recent within the last 5 years)
* Prior administration of anthracyclines is acceptable if therapy was completed > 6 months prior to study enrollment
* Patients that are receiving or have received chemotherapy regimens are allowed
* Able to hold breath for 10 seconds
* Prior cancers allowed if no evidence of disease in last 5 years
* Eastern Cooperative Oncology Group (ECOG) 0 or 1

Exclusion Criteria:

* Prior use of lipid-lowering therapy within the last 6 months
* Current postmenopausal hormone-replacement therapy
* Uncontrolled hypertension (systolic blood pressure >190 mm Hg or diastolic blood pressure >100 mm Hg)
* Scheduled to receive neoadjuvant chemotherapy with an anthracycline
* No active liver disease allowed
* Uncontrolled hypothyroidism
* Recent history (within past 3 years) of alcohol or drug abuse, inflammatory conditions such as lupus or inflammatory bowel disease, use of immunosuppressant agents, or another medical condition that might compromise safety or the successful completion of the study.
* Patients with ferromagnetic cerebral aneurysm clips or other intraorbital/intracranial metal;pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices.
* Unstable angina; significant ventricular arrhythmias (>20 premature ventricular complexes (PVCs)/min due to gating difficulty) atrial fibrillation with uncontrolled ventricular response; coronary artery disease; acute myocardial infarction within 28 days
* Current use of Cytochrome P450 (CYP3A4) inhibitors. These include Clarithromycin, HIV protease inhibitors, Itraconazole, grapefruit juice, Cyclosporine, Rifampin or Digoxin
* Current or history of hepatic dysfunction
* Unable to provide informed consent
* Claustrophobia
* Planning to move within 24 months of trial enrollment
* Pregnant or breast-feeding

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hundley, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (51):
- United States (51):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Mission Hospital, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin

REFERENCES:
- [Derived] Grizzard PJ, O'Connell NS, Rapp SR, Olson KC, Bellissimo MP, Hughes AN, Ladd AC, Weaver KE, Wagner LI, Ruddy KJ, Ky B, D'Agostino RB, Hundley WG. Preserved Cognitive Function After Statin Administration During Cancer Treatment With Doxorubicin: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2538325. doi: 10.1001/jamanetworkopen.2025.38325. PMID 41118164
- [Derived] Sutton AL, O'Connell NS, Lucas AR, Olson KC, Reding KW, Sheppard VB, Ky B, Ruddy KJ, Weaver KE, Hundley WG. Socioeconomic status and left ventricular ejection fraction decline in breast cancer survivors following receipt of doxorubicin (PREVENT WF-98213). Cardiooncology. 2025 Feb 5;11(1):11. doi: 10.1186/s40959-025-00311-y. PMID 39910652
- [Derived] Hundley WG, D'Agostino R Jr, Crotts T, Craver K, Hackney MH, Jordan JH, Ky B, Wagner LI, Herrington DM, Yeboah J, Reding KW, Ladd AC, Rapp SR, Russo S, O'Connell N, Weaver KE, Dressler EV, Ge Y, Melin SA, Gudena V, Lesser GJ. Statins and Left Ventricular Ejection Fraction Following Doxorubicin Treatment. NEJM Evid. 2022 Sep;1(9):10.1056/evidoa2200097. doi: 10.1056/evidoa2200097. Epub 2022 Aug 18. PMID 36908314

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No reason for exclusion prior to randomization.
Period: Overall Study
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Started | 139 | 140
Completed Baseline (Defined as having labs done at that time point.) | 136 | 139
Completed 6 Month Visit (Defined as having labs done at that time point.) | 122 | 126
Completed (Defined as having labs done at that time point.) | 100 | 105
Not Completed | 39 | 35
Not completed — Death | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 31 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo | Total
Number analyzed (Participants) | 139 | 140 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.5) | 49.4 (11.5) | 49.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 127 | 256
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 134 | 136 | 270
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 16 | 22 | 38
  White | 115 | 116 | 231
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Medicare [Count of Participants; unit: Participants] — Number of participants on Medicare. Insurance categories are check all that apply, participants could report more than 1 insurance type.
  Participants | 16 | 10 | 26
Medicaid [Count of Participants; unit: Participants] — Number of participants on Medicaid. Insurance categories are check all that apply, participants could report more than 1 insurance type.
  Participants | 10 | 11 | 21
Private Insurance [Count of Participants; unit: Participants] — Number of participants on private health insurance. Insurance categories are check all that apply, participants could report more than 1 insurance type.
  Participants | 112 | 121 | 233
No Health Insurance [Count of Participants; unit: Participants] — Number of participants reporting having no health insurance
  Participants | 6 | 1 | 7
Cancer Type [Count of Participants; unit: Participants] — Defined as lymphoma or breast cancer (those were the only two types eligible for this trial).
  Participants
    Lymphoma | 20 | 21 | 41
    Breast Cancer | 119 | 119 | 238
Cancer Stage [Count of Participants; unit: Participants] — Clinical staging is based on the results of tests done before surgery, which may include physical examinations, ultrasound, and MRI scans. Cancer stages range from 1-4. The higher the number, the larger the cancer tumor and the more it has spread to nearby tissues. Stage 4 has spread to distant parts of the body. Higher stages are associated with worse prognosis.
  Participants
    Stage 1 | 24 | 22 | 46
    Stage 2 | 77 | 77 | 154
    Stage 3 | 34 | 40 | 74
    Stage 4 | 4 | 1 | 5
Marital Status [Count of Participants; unit: Participants]
  Single, Never Married | 23 | 15 | 38
  Married | 82 | 84 | 166
  Living in a married like relationship | 4 | 8 | 12
  Separated or Divorced | 23 | 25 | 48
  Widowed | 3 | 3 | 6
  Unknown | 4 | 5 | 9
Education [Count of Participants; unit: Participants] — Self reported highest level of education.
  Participants
    Grades 1-8 | 2 | 0 | 2
    Grades 9-11 | 3 | 3 | 6
    High School/GED | 28 | 16 | 44
    Vocational/trading school | 4 | 6 | 10
    Some College/Assoicates | 27 | 49 | 76
    College Degree (Bachelors) | 36 | 32 | 68
    Some post college | 6 | 7 | 13
    Masters degree | 21 | 16 | 37
    Doctoral degree | 1 | 3 | 4
    Unknown | 11 | 8 | 19
Income [Count of Participants; unit: Participants] — Self reported annual income.
  Participants
    Less than $10,000 | 11 | 6 | 17
    $10,000-$20,000 | 14 | 12 | 26
    $20,000-$35,000 | 12 | 19 | 31
    $35,000-$50,000 | 15 | 12 | 27
    $50,000-$75,000 | 27 | 30 | 57
    $75,000-$100,000 | 11 | 16 | 27
    $100,000-$150,000 | 10 | 10 | 20
    More than $150,000 | 7 | 5 | 12
    Unknown | 32 | 30 | 62
Job Status [Count of Participants; unit: Participants]
  Not currently working | 16 | 14 | 30
  Retired | 15 | 14 | 29
  Homemaker | 10 | 4 | 14
  Employed | 83 | 95 | 178
  Disabled, unable to work | 7 | 7 | 14
  Other | 5 | 3 | 8
  Unknown | 3 | 3 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — kg/m^2
  kg/m^2 | 29 (6.43) | 31 (7.4) | 30 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: 24 month estimated values of clinical measurements obtained from Cardiac MRI left ventricular ejection fraction by group. Linear model adjusts for baseline value and group assignment and multiple imputation was utilized for missing data.
Time Frame: 24 months
Population: All those with baseline and 24 month cardiac MRI (multiple imputation utilized for missing data).
Measure: Least Squares Mean (Standard Error); unit: percent ejected from LV per heartbeat
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
percent ejected from LV per heartbeat | 58.1 (0.555) | 57.9 (0.560)
Statistical Analysis 1: Comparison: Arm 1 - Atorvastatin vs Arm 2 - Placebo; Linear models adjusting for baseline values and utilized multiple imputation for missing data; Test type: Superiority — Power described in protocol; p = 0.84, ANCOVA; Adjusted for multiple imputation of missing data; Mean Difference (Net) = 0.1608, Standard Error of Mean 0.7787

2. Secondary Outcome: End Diastolic Volume
Description: 24 month estimated values of clinical measurements obtained from Cardiac MRI End Diastolic Volume by group. Linear model adjusts for baseline value and group assignment and multiple imputation was utilized for missing data.
Time Frame: 24 months
Population: All those with baseline and 24 month cardiac MRI (multiple imputation utilized for missing data).
Measure: Least Squares Mean (Standard Error); unit: milliliters of blood
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
milliliters of blood | 123 (2.06) | 125 (2.01)

3. Secondary Outcome: End Systolic Volume
Description: 24 month estimated values of clinical measurements obtained from Cardiac MRI End Systolic Volume by group. Linear model adjusts for baseline value and group assignment and multiple imputation was utilized for missing data.
Time Frame: 24 months
Population: All those with baseline and 24 month cardiac MRI (multiple imputation utilized for missing data).
Measure: Least Squares Mean (Standard Error); unit: milliliters of blood
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
milliliters of blood | 51.8 (1.27) | 52.9 (1.25)

4. Secondary Outcome: Stroke Volume
Description: 24 month estimated values of clinical measurements obtained from Cardiac MRI Stroke Volume by group. Linear model adjusts for baseline value and group assignment and multiple imputation was utilized for missing data.
Time Frame: 24 months
Population: All those with baseline and 24 month cardiac MRI (multiple imputation utilized for missing data).
Measure: Least Squares Mean (Standard Error); unit: milliliters per minute
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
milliliters per minute | 71 (1.58) | 72.2 (1.50)

5. Secondary Outcome: Left Ventricular (LV) Mass
Description: 24 month estimated values of clinical measurements obtained from Cardiac MRI left ventricular mass by group. Linear model adjusts for baseline value and group assignment and multiple imputation was utilized for missing data.
Time Frame: 24 months
Population: All those with baseline and 24 month cardiac MRI (multiple imputation utilized for missing data).
Measure: Least Squares Mean (Standard Error); unit: gram per meter squared
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
gram per meter squared | 88.4 (1.68) | 87.5 (1.65)

6. Secondary Outcome: Pulse Wave Velocity
Description: 24 month estimated values of clinical measurements obtained from Cardiac MRI pulse wave velocity by group. Linear model adjusts for baseline value and group assignment and multiple imputation was utilized for missing data.
Time Frame: 24 months
Population: All those with baseline and 24 month cardiac MRI (multiple imputation utilized for missing data).
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
m/s | 5.73 (0.247) | 5.51 (0.24)

7. Secondary Outcome: Hopkins Verbal Learning Test (HVLT) Total Recall
Description: 24 month estimated values Hopkins Verbal Learning test (HVLT) total recall by group. Linear model adjusts for baseline value and group assignment. No missing imputation performed. Ranges from 0 to 36 and higher numbers reflect better recall.
Time Frame: 24 months
Population: Those with data available at baseline and 24 months.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
score on a scale | 28.5 (0.518) | 27.5 (0.503)

8. Secondary Outcome: Controlled Oral Word Association (COWA)
Description: 24 month estimated values Controlled Oral Word Association (COWA) by group. Linear model adjusts for baseline value and group assignment. No missing imputation performed. The COWA uses the three letter set of C, F, and L to assess phonemic fluency. Individuals are given 1 min to name as many words as possible beginning with one of the letters. The procedure is then repeated for the remaining two letters. Ranges from 0 to the total number of correct words that begin with one of the letters in the set. There is no ceiling of a maximum score. Higher numbers reflect better verbal fluency.
Time Frame: 24 months
Population: Those with data available at baseline and 24 months.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
score on a scale | 41.6 (1.07) | 44.7 (1.06)

9. Secondary Outcome: Patient-reported Outcomes Measurement (PROMIS) Questionnaire - Applied Cognition - General Concerns - Short Form 4a
Description: Patient reported quality of life outcomes obtained from patient-reported outcomes measurement (PROMIS) questionnaire - Applied Cognition - General Concerns - Short Form 4a . Scores range from 4-20 and then adjusted by t-scores ranging from 30.1-63.8. Higher scores reflect better cognition. Linear models include baseline assessment and group and multiple imputation was utilized.
Time Frame: 24 months
Population: Those with baseline and 24 month assessment completed. Multiple imputation was utilized for missing data.
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
t-score | 45.57 (1.1) | 46.55 (1.14)

10. Secondary Outcome: Patient-reported Outcomes Measurement (PROMIS) Questionnaire - Fatigue Short Form 41
Description: Patient reported quality of life outcomes obtained from patient-reported outcomes measurement (PROMIS) questionnaire - Fatigue Short Form 41. Scores range from 4-20 and then adjusted by t-scores ranging from 33.7-75.8. Higher scores reflect worse fatigue. Linear models include baseline assessment and group and multiple imputation was utilized.
Time Frame: 24 months
Population: Those with baseline and 24 month assessment completed. Multiple imputation was utilized for missing data.
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
Number analyzed (Participants) | 136 | 139
t-score | 48.17 (1.08) | 49.29 (1.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire trial and up to 30 days post-completion of statin or placebo (approximately 25 months)
Description: Serious Adverse Event reporting begins after the informed consent is signed. Serious Adverse Events occurring within 30 days of study completion must be reported via FDA Form 3500 (MedWatch).
Arm/Group | Arm 1 - Atorvastatin | Arm 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 3/139 | 1/140
Serious Adverse Events (participants affected / at risk) | 17/139 | 18/140
Other Adverse Events (participants affected / at risk) | 0/139 | 0/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Atorvastatin (N=139) | Arm 2 - Placebo (N=140)
Febrile neutropenia (Infections and infestations) | 3 | 7
Hospitalization for Reconstructive Surgery (Surgical and medical procedures) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Herpes simplex reactivation (Infections and infestations) | 1 | 1
Decreased neutophils (Investigations) | 1 | 1
White blood cells decreased (Blood and lymphatic system disorders) | 0 | 1
Cardiac Disorder (Cardiac disorders) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back Pain (Injury, poisoning and procedural complications) | 1 | 0
Breast Infection (Infections and infestations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Nervous System Disorder (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT01988571/Prot_SAP_001.pdf
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT01988571/ICF_000.pdf